CLINICAL TRIAL: NCT05855044
Title: Efficacy of External Application of Rosemary Oil in Patients With Chemotherapy-Induced Peripheral Neuropathy - a Monocentre, Single-arm Non-controlled Feasibility Study to Assess the Feasibility of Evaluating Topical Applications in CIPN
Brief Title: Efficacy of External Application of Rosemary Oil in Patients With Chemotherapy-Induced Peripheral Neuropathy: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPN_01
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN)
Keywords: Chemotherapy-induced peripheral neuropathy; Oncological patients; Cancer; Chemotherapy; Rosemary oil
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rosemary oil (Experimental)
  Interventions: Other: Rosemary oil application

INTERVENTIONS:
Other: Rosemary oil application — Application of Rosemary oil (10%) to both hands and both feet once a day for 24 weeks

SUMMARY:
Chemotherapy can cause sensory disorders in the hands and feet called peripheral neuropathy. Typical symptoms are pain, loss of sensation, tingling, numbness, and gait disturbances, which worsen patients' quality of life and increase the risk of falls. Little is known about the effect of rosemary oil (applied to hands and feet) on the symptoms of neuropathy. The present study is a feasibility study to see if it is possible to conduct a clinical trial in patients diagnosed with cancer and receiving chemotherapy who report peripheral neuropathy and apply rosemary oil to their hands and feet.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most common severe dose-limiting side effects that accompany treatment with different chemotherapeutic agents. Patients with CIPN often experience a reduction in quality of life and an increase in fall risk due to symptoms such as pain, sensory loss, paresthesia (tingling, numbness), and gait disturbances. Treatment of CIPN is based on pharmacotherapy, which may in turn cause side effects such as nausea, dizziness, fatigue and others. In addition, various approaches from integrative medicine are used, e.g. acupuncture, touch therapies, mind-body medicine, dietary supplements, and aromatherapy. Little is known about the effect of rosemary oil, applied to hands and feet, on CIPN. The present study is a feasibility study to determine the feasibility of a future clinical trial to investigate the efficacy of topical application of rosemary oil in cancer patients undergoing chemotherapy who develop CIPN.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 years or older
* Cancer diagnosis
* Assignment to neurotoxic chemotherapy that has not yet started at the time of enrolment
* Intact, irritation-free skin on the hands and feet
* No history of neuropathic pain

Exclusion Criteria:

* Neurorelevant comorbidities such as diabetes or alcohol abuse
* Use of medication for neuropathy such as gabapentin, pregabalin, venlafaxine or duloxetine
* Other relevant treatments for CIPN during the study
* Insufficient knowledge of the German language
* History of rosemary oil allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Participation rate | When participation in the study is offered, before start of chemotherapy and rosemary oil application
  Participation rate in relation to all eligible patients and the reasons for non-participation. Reasons for refusal to participate in the study will be recorded.

SECONDARY OUTCOMES:
Rate of fully completed EORTC QLQ-CIPN20 questionnaires | Before start of chemotherapy and rosemary oil application (baseline), then weekly for 24 weeks
  The rate of fully completed EORTC QLQ-CIPN20 questionnaires in relation to incomplete questionnaires and reasons for missing data. EORTC QLQ-CIPN20 is used to measure the severity of CIPN pain and functional symptoms. It includes 20 items in three subscales to evaluate sensory (9 items), autonomic (3 items) and motor (8 items) symptoms and function. Each item is rated on a four-point Likert scale from 1 (not at all) to 4 (very much). Scores are summed up to a total score, which is linearly converted to a scale of 0-100 (a high score means more symptoms and pain).
Efficacy of rosemary oil according to EORTC QLQ-CIPN20 questionnaire | Before start of chemotherapy and rosemary oil application (baseline), then weekly for 24 weeks
  Efficacy of rosemary oil in order to obtain a basis for a sample size calculation in a follow-up study. Effect of rosemary oil application will be measured using the EORTC QLQ-CIPN20 questionnaire. EORTC QLQ-CIPN20 is used to measure the severity of CIPN pain and functional symptoms. It includes 20 items in three subscales to evaluate sensory (9 items), autonomic (3 items) and motor (8 items) symptoms and function. Each item is rated on a four-point Likert scale from 1 (not at all) to 4 (very much). Scores are summed up to a total score, which is linearly converted to a scale of 0-100 (a high score means more symptoms and pain).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr., Study Director — ARCIM Institute Academic Research in Complementary and Integrative Medicine
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available, in addition to study protocol and informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.